CLINICAL TRIAL: NCT05106790
Title: Efficacy of mHealth and Education-led Peer Counseling of Patients With Hypertension and Coronary Artery Disease: a Double-blinded Pragmatic Randomized Control Trial With Factorial Design, Pakistan
Brief Title: A Factorial Approach to Improve Treatment Adherence and Systolic Blood Pressure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD studentship, Universiti Putra Malaysia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: APUTRA
Record Dates: First submitted 2021-10-23; First posted 2021-11-04 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2022-05

CONDITIONS: Treatment Adherence and Compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: It's a 12-month factorial design, intention-to-treat, four-arm, double-blinded, multicentre, pragmatic randomized controlled trial with an intervention to assess the efficacy of mHealth and education support with peer counseling to improve treatment adherence and lower systolic blood pressure in hypertensive patients in three teaching hospitals in Lahore, Pakistan.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard care arm (No Intervention): The first group will be on standard care as usually being practiced in hospitals.
- Ed-counseling arm (Active Comparator): The second group will receive monthly educational support ( booklets) with peer counseling sessions in addition to standard care.
  Interventions: Behavioral: Educational support with peer counseling
- mHealth (Active Comparator): The third group will receive daily written and voice reminders, and once weekly an education-led video in addition to standard care.
  Interventions: Behavioral: mHealth intervention
- Combined arm (Active Comparator): The fourth group will receive educational support (booklets)and counseling sessions every month, daily written and voice reminders, and once weekly an education-led video in addition to standard care.
  Interventions: Behavioral: mHealth intervention and Educational support with peer counseling

INTERVENTIONS:
Behavioral: Educational support with peer counseling — This group will receive peer counseling therapy sessions will be led by doctors who specialize in hypertension. Patients and their families will be the focus of the sessions. Face-to-face sessions will take roughly 25-30 minutes. Patients will receive spoken and written instructions based on their abilities during these sessions. The counseling sessions are geared toward overcoming both general and personal obstacles. The educational component will be delivered through smart booklets. Information on hypertension, blood pressure self-monitoring, and frequent systolic blood pressure (SBP) tests, as well as body weight and serum cholesterol values, are included in the instructional support. Food control, exercise therapy, and hypertension problems and their management will also be explored as non-pharmacological therapeutic approaches.
  Arms: Ed-counseling arm
Behavioral: mHealth intervention — This group will receive mHealth intervention will include daily written and voice messages, and once weekly an educational-led video. This intervention module will be delivered through "WhatsApp".
  Arms: mHealth
Behavioral: mHealth intervention and Educational support with peer counseling — This group will receive both Educational support (Smart booklets) with peer counseling sessions on a monthly basis and mHealth intervention will include daily written and voice reminders, and once weekly an educational led video.
  Arms: Combined arm

SUMMARY:
In Pakistan, poor medication adherence is a key operational factor in the prevalence of uncontrolled hypertension. Mobile phone treatments based on technology are at the forefront and are a reasonably low-cost strategy for combating the latest health concerns associated with poor adherence. On the other hand, conservative approaches to counseling are also found effective. This study will look at how a mHealth-based strategy and an educational-led peer counseling intervention can help hypertensive patients with coronary artery disease lower their systolic blood pressure.

DETAILED DESCRIPTION:
In Pakistan, hypertension is a serious public health concern. Hypertension affects 18.9% of teenagers over the age of 15 and 33% of adults over the age of 45; however, only around 3% of hypertensive individuals have their blood pressure regulated to 140/90 mm Hg or lower. The majority of hypertensive patients are found to have blood pressure that is out of control. The majority of those undergoing therapies were judged to be non-compliant. According to the study, adherence to cardiac medications ranged from 27 to 77 percent, while adherence to stroke medications was around 68 percent. According to a recent study, 37.7% of patients did not take their antihypertensive medication as advised.

Interventions to help hypertensive patients in controlling blood pressure show potential to alter their behavior and lead to better outcomes, but delivering them at a cheap cost is difficult. Although evidence is scarce, several trials examining clinical interventions utilizing conventional health education support while others employing a mobile health strategy, both showed significant results. For a low-resource country, we built cost-effective models that are integrated with clinical care for patients with hypertension. The goal of this trial is to assess the effectiveness of mHealth intervention with clinical educational support and educational support with peer counseling to improve blood pressure control in hypertensive patients when compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Participants with age 21 to 70 years
* Participants who have been registered as hypertensive with comorbidity of coronary artery disease in the Outpatient Departments (OPDs) of one of the three public teaching hospitals in Lahore, for at least last one month
* Participants on antihypertensive drugs
* The participants with stable coronary artery disease who are treated in an outpatient setting
* Participants who are willing to sign a written informed consent form, must have a smartphone with the WhatsApp application installed and be able to read Urdu/English.
* Participants with smartphones and have internet access

Exclusion Criteria:

Participants who suffer from some type of malignancy and require adjustment of drugs

* Participants with any biological condition that makes it difficult for them to read write, communicate or hear phone calls
* Participants in hypertensive emergency blood pressure >220/120 mmHg
* Participants with pregnancy(self-reporting)
* Participants in their period of lactation

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1440 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in systolic blood pressure (SBP) | 12- month from baseline
  The primary outcome is a change in systolic blood pressure (SBP) of participants at 0, 6, and 12 months. The blood pressure will be recorded by sphygmomanometer used was calibrated upper-arm electronic sphygmomanometer (OMRON HEM-7200, OMRON Corporation, Dalian). Two separate readings will be taken within 5 min, and the average measurement will be the final. If the difference between the two measurements will be more than 5mmHg, then a third recording will be done and the average is considered.
Proportion of participants achieving blood pressure < 140/90 mmHg | 12- month from baseline
  The proportion of participants achieving the control blood pressure < 140/90 mmHg
Proportion of participants attending scheduled clinic appointments | 12- month from baseline
  The proportion of participants attending scheduled clinic appointments

SECONDARY OUTCOMES:
Measuring quality of life | 12- month from baseline
  To measure the health-related quality of life at baseline, three-month, and 12-month post-intervention, EuroQol 5-Dimension- 3-level will be used. The European quality of life scale (EQ-5D-3L) has five dimensions and three levels. Each of the five dimensions comprising the EQ-5D descriptive system is divided into three levels of perceived problems: LEVEL 1: indicating no problem LEVEL 2: indicating some problems LEVEL 3: indicating extreme problems, 1 (perfect health), with higher scores indicating higher health utility.
  2- On a 20 cm vertical visual analog scale, the EQ-VAS captures the patient's self-rated health, with two unique endpoints such as "Best imaginable health condition" for a score of 100 and "Worst imaginable health state" for a score of 0.

OTHER OUTCOMES:
Change in medication adherence to antihypertensive treatment | 12- month from baseline
  1. The secondary outcome is the change in medication adherence to antihypertensive treatment. Using the "pills taken over a certain period, divided by pills prescribed for that specific period", the primary outcome will be measured.it will be self-reporting. A cut-off value of 80% has been established from previous literature. Non-adherents will make up less than 80% of the population, while adherents will make up more than 80%.
  2. The SEAMS is a 13-item questionnaire that has three-point responses. The score for the 13-item scale ranges from 13 to 39. Higher scores show better levels of self-efficacy for medication adherence and vice versa.

CONTACTS AND LOCATIONS:
Overall Officials: Arshed MUHAMMAD, Principal Investigator — UPM
Locations (6):
- Pakistan (6):
  - Victoria Hospital, Bahawalpur, Punjab Province
  - Sheikh Zayed Hospital Rahim Yar Khan, Rahim Yar Khan, Punjab Province
  - Jinnah Hospital, Lahore
  - Punjab Institute of Cardiology, Lahore
  - Rehmatul-lil-Almeen Institute of Cardiology, Lahore
  - Sheikh Zayed, Hospital, Lahore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NCD Risk Factor Collaboration (NCD-RisC). Worldwide trends in blood pressure from 1975 to 2015: a pooled analysis of 1479 population-based measurement studies with 19.1 million participants. Lancet. 2017 Jan 7;389(10064):37-55. doi: 10.1016/S0140-6736(16)31919-5. Epub 2016 Nov 16. PMID 27863813
- [Background] Lewington S, Clarke R, Qizilbash N, Peto R, Collins R; Prospective Studies Collaboration. Age-specific relevance of usual blood pressure to vascular mortality: a meta-analysis of individual data for one million adults in 61 prospective studies. Lancet. 2002 Dec 14;360(9349):1903-13. doi: 10.1016/s0140-6736(02)11911-8. PMID 12493255
- [Background] NIPS/Pakistan and ICF NI of PS-. Pakistan Demographic and Health Survey 2017-18. 2019 [cited 4 Jan 2021]. Available: https://dhsprogram.com/publications/publication-fr354-dhs-final-reports.cfm
- [Background] Mahmood S, Jalal Z, Hadi MA, Orooj H, Shah KU. Non-Adherence to Prescribed Antihypertensives in Primary, Secondary and Tertiary Healthcare Settings in Islamabad, Pakistan: A Cross-Sectional Study. Patient Prefer Adherence. 2020 Jan 14;14:73-85. doi: 10.2147/PPA.S235517. eCollection 2020. PMID 32021119
- [Background] Zhai P, Hayat K, Ji W, Li Q, Shi L, Atif N, Xu S, Li P, Du Q, Fang Y. Efficacy of Text Messaging and Personal Consultation by Pharmacy Students Among Adults With Hypertension: Randomized Controlled Trial. J Med Internet Res. 2020 May 20;22(5):e16019. doi: 10.2196/16019. PMID 32432556
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Bhide A, Shah PS, Acharya G. A simplified guide to randomized controlled trials. Acta Obstet Gynecol Scand. 2018 Apr;97(4):380-387. doi: 10.1111/aogs.13309. Epub 2018 Feb 27. PMID 29377058
- [Background] Risser J, Jacobson TA, Kripalani S. Development and psychometric evaluation of the Self-efficacy for Appropriate Medication Use Scale (SEAMS) in low-literacy patients with chronic disease. J Nurs Meas. 2007;15(3):203-19. doi: 10.1891/106137407783095757. PMID 18232619
- [Background] Strobl J, Cave E, Walley T. Data protection legislation: interpretation and barriers to research. BMJ. 2000 Oct 7;321(7265):890-2. doi: 10.1136/bmj.321.7265.890. No abstract available. PMID 11021874
- [Background] Del Re AC, Maisel NC, Blodgett JC, Finney JW. Intention-to-treat analyses and missing data approaches in pharmacotherapy trials for alcohol use disorders. BMJ Open. 2013 Nov 12;3(11):e003464. doi: 10.1136/bmjopen-2013-003464. PMID 24227870
- [Background] Montgomery AA, Peters TJ, Little P. Design, analysis and presentation of factorial randomised controlled trials. BMC Med Res Methodol. 2003 Nov 24;3:26. doi: 10.1186/1471-2288-3-26. PMID 14633287
- [Background] Whelan DB, Dainty K, Chahal J. Efficient designs: factorial randomized trials. J Bone Joint Surg Am. 2012 Jul 18;94 Suppl 1:34-8. doi: 10.2106/JBJS.L.00243. PMID 22810445